CLINICAL TRIAL: NCT02098135
Title: Phase 1 Study of a Home Therapy and Assessment for Patients With Arm Impairments
Brief Title: ArmeoSenso - Home Therapy and Assessment for Patients With Arm Impairments Based on Wearable Movement Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0182
Record Dates: First submitted 2014-03-06; First posted 2014-03-27 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Stroke; Spinal Cord Injury
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ArmeoSenso (Experimental): The ArmeoSenso system is an easy to set up and use upper limb rehabilitation system for the home environment. It consists of a motion capture system based on wearable sensors in combination with a personal computer as well as a therapy software that provides an ergonomic user interface, therapy games and automated assessments.
  Interventions: Device: ArmeoSenso

INTERVENTIONS:
Device: ArmeoSenso — Virtual realty therapy with a touchscreen computer and movement sensors, over 42 days.

SUMMARY:
stroke, spinal cord injury, rehabilitation, home therapy, upper limb, arm, virtual reality, interia sensor,

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* 18 years old
* Stroke or spinal cord injury in prehistory
* Motor deficits of the upper limb (s)
* Lifting the paretic arm against gravity possible AND
* Minimum amount of movement in the horizontal plane of 20 x 20 cm
* Ability and willingness to participate in the study

Exclusion criteria:

* Severe aphasia
* Severe dementia
* Severe depression
* Relevant restriction of vision, which can not be compensated by aids (eg hemianopia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Numbers of participant which can perform the ArmeoSenso - training. | 42 days

SECONDARY OUTCOMES:
Improvement in the Arm function | 42 days
  WMFT (Wolf Motor Function Test), FMA-UL (Fugl-Meyer Assessment - Upper Limb), GRASSP (Graded and Redefined Assessment of Strength, Sensibility and Prehension)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Luft, Prof MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Divison of Neurology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Wittmann F, Held JP, Lambercy O, Starkey ML, Curt A, Hover R, Gassert R, Luft AR, Gonzenbach RR. Self-directed arm therapy at home after stroke with a sensor-based virtual reality training system. J Neuroeng Rehabil. 2016 Aug 11;13(1):75. doi: 10.1186/s12984-016-0182-1. PMID 27515583